CLINICAL TRIAL: NCT05970081
Title: Effectiveness and Safety of Implantable Intrathecal Systems for the Treatment of Chronic Refractory Pain in Spain: Prospective Multicenter Study From the Spanish Pain Society Registry (INTRATHECAL-RENASED)
Brief Title: Effectiveness and Safety of Implantable Intrathecal Systems for Refractory Pain in Spain (INTRATHECAL-RENASED)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sociedad Espanola del Dolor (Other)
Responsible Party: Sponsor
Other Study IDs: 5215
Record Dates: First submitted 2023-07-24; First posted 2023-08-01 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2023-09

CONDITIONS: Refractory Pain
Keywords: Intrathecal Drug Delivery; Implantable Infusion Pump; Refractory Pain
MeSH Terms: conditions — Pain, Intractable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Refractory pain is a prevalent condition that negatively affects patients' quality of life. Intrathecal implantable systems have been proposed as a treatment option for refractory pain. However, real-world data on the effectiveness and safety of these therapies in Spain are scarce. This study aims to obtain real-world data on the effectiveness and safety of intrathecal implantable systems for refractory pain treatment in Spain.

DETAILED DESCRIPTION:
All Spanish hospitals that implant intrathecal systems for refractory pain will be invited to participate in the study. Patients will be recruited before the procedure, and before providing data to the registry, the study will be explained to them, and they will sign an informed consent form. Demographic data related to the pathology and procedure will be collected. Follow-up will be conducted at three and twelve months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Chronic refractory pain patients candidates for treatment with an implantable neurostimulation system.
* Accept to participate in the study and sign informed consent.

Exclusion Criteria:

* Patients in whom it would be difficult to complete follow-up.
* Insufficient understanding of the Spanish language.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with refractory pain who are candidates for treatment with an implantable intrathecal infusion system.
Sampling Method: Non-Probability Sample
Enrollment: 504 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with at least 50 percent pain relief in the area of their predominant pain at one year | Twelve months
  Percentage of patients who experience a reduction of at least 50 percent in the intensity of their predominant pain compared to the initial value, assessed twelve months after the implantation of the intrathecal drug delivery system. Pain intensity will be measured using an 11-point Numeric Pain Rating Scale (NPRS), with a range from 0 (no pain) to 10 (maximum pain possible)

SECONDARY OUTCOMES:
Percentage of patients with at least 50 percent pain relief in the area of their predominant pain at three months | Three months
  Percentage of patients who experience a reduction of at least 50 percent in the intensity of their predominant pain compared to the initial value, assessed three months after the implantation of the implantable intrathecal system. Pain intensity will be measured using an 11-point Numeric Pain Rating Scale (NPRS), with a range from 0 (no pain) to 10 (maximum pain possible)
Percentage of patients with at least 50 percent pain relief in the area of their non-predominant pain at one year | Twelve months
  Percentage of patients who experience a reduction of at least 50 percent in the intensity of their non-predominant pain compared to the initial value, assessed twelve months after the implantation of the intrathecal drug delivery system. Pain intensity will be measured using an 11-point Numeric Pain Rating Scale (NPRS), with a range from 0 (no pain) to 10 (maximum pain possible)
Compared change from baseline on health-related quality of life scores (EQ Index) | Three and twelve months
  The impact of the treatment on the patient's health-related quality of life will be evaluated using the EQ-5D-5L questionnaire at three and twelve months after implantation. The EQ-5D-5L assesses quality of life across five domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each domain is scored on a scale of 1 (no problems) to 5 (extreme problems), generating a 5-digit code that corresponds to the patient's health status.
Patient Global Impression of Improvement (PGI-I) | Three and twelve months
  Assessment of clinical global impression of improvement using the PGI-I scale at three and twelve months after implantation of the intrathecal drug delivery system. The PGI-I score ranges from 1 (Very much better) through to 7 (Very much worse). The lower the score, the better the improvement.
Patient Satisfaction | Three and twelve months
  Percentage of implanted subjects satisfied with the treatment at three and twelve months after the implantation of the intrathecal drug delivery system. Defined as indicating: "since the start of the therapy has the pain improved? yes/no", "Are you satisfied with the treatment?" yes/no or "would you agree to the treatment again?" yes/no
Number of Adverse Events as a Measure of Safety | Three and twelve months
  Number and percentage of patients with adverse effects related to therapy at three and twelve months after implantation of the intrathecal drug delivery system.

CONTACTS AND LOCATIONS:
Locations (9):
- Spain (9):
  - Hospital Regional Univeristario de Málaga, Málaga, Andalusia
  - Hospital Universitari Son Espases, Palma de Mallorca, Balearic Island
  - Hospital Universitario de Navarra, Pamplona, Navarre
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Madrid
  - Complejo Hospitalario Universitario de Cartagena, Murcia
  - Complexo Hospitalario Univeritario de Ourense, Ourense
  - Hospital Universitari i Politècnic La Fe, Valencia